CLINICAL TRIAL: NCT04538846
Title: Culinary Art Therapy Group for Adults With Eating Disorders: Assessment of Influence on Thinking, Patterns and Behaviour Related to Food.
Brief Title: Culinary Art Therapy Group for Adults With Eating Disorders.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Principal Investigator, Adi Schleyer, Dr., Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0482-20-HMO
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Eating Disorders; Behavior, Eating; Relationship, Family; Cognitive Change
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Quasi-Experimental Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culinary Art Therapy Group (Experimental): Patients with eating disorders that will participate in a weekly session of culinary art therapy group.
  Interventions: Other: Culinary art therapy
- No Culinary Art Therapy Intervention (No Intervention): Patients with eating disorders that are not scheduled to come to the outpatients ward on the day of intervention.

INTERVENTIONS:
Other: Culinary art therapy — Culinary art therapy is a novel approach which broadly perceives food and cooking as enabling participants to explore needs, patterns and relationships and facilitate therapeutic processes.
  Arms: Culinary Art Therapy Group

SUMMARY:
The study will assess the influence of culinary art therapy group (a new therapeutic tool) for adults with eating disorders. It will assess changes in thinking patterns and behavioural patterns associated with food and eating.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of eating disorder
* Body Mass Index (BMI) > 15

Exclusion Criteria:

* No active participation in three group sessions
* Refusal to take an active part in the sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Eating Attitudes Test (EAT-26) | 3 months
  This is a screening measure to help determine whether a person might have an eating disorder that needs professional attention. This screening measure is not designed to make a diagnosis of an eating disorder or take the place of a professional consultation.
Eating & Meal Preparation Skills Questionnaire (EMPSA) | 3 months
  The EMPSA is a 12-item self-report assessment tool designed to measure eating disordered clients' perceived ability and motivation to perform 12 eating and meal preparation tasks.
Rosenberg Self-Esteem Scale (RSES) | 3 months
  The Rosenberg Self-Esteem Scale (RSES) assesses global self-esteem and sense of self-worthiness.

SECONDARY OUTCOMES:
Assessment of Communication and Interaction Skills (ACIS) | 3 months
  The ACIS is an observational assessment that gathers data on communication and interaction skills. Three domains, physicality, information exchange, and relations, are used to describe different aspects of communication and interaction. The ACIS gathers data on skill as it is exhibited during performance in an occupational form and/or within a social group.
Individual semi-structured interview | 3 months
  Interviews aimed to allow each participant to relate to his or her own experience in a more independent and possibly safer setting.

CONTACTS AND LOCATIONS:
Overall Officials: Adi Stern, Dr., Principal Investigator — University of Haifa
Locations (1):
- Eating disorders outpatients department, Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No